CLINICAL TRIAL: NCT01350388
Title: Effects of Febuxostat on Adipokines and Kidney Disease in Diabetic Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Srinvasan Beddhu, Srinivasan Beddhu, MD Associate Professor of Medicine, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB_00044016
Record Dates: First submitted 2011-04-20; First posted 2011-05-09 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Kidney Disease; Diabetes
Keywords: Chronic Kidney Disease; Diabetes; Febuxostat; Inflammation; Hyperuricemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Inflammation; Hyperuricemia | interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Febuxostat (Active Comparator): 80 mg/day of febuxostat for 24 weeks
  Interventions: Drug: Febuxostat
- Placebo (Placebo Comparator): 1 placebo tablet per day for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Febuxostat — 80 mg/day of febuxostat for 24 weeks
  Other Names: Uloric
  Arms: Febuxostat
Drug: Placebo — 1 placebo tablet per day for 24 weeks
  Arms: Placebo

SUMMARY:
Hyperuricemia is emerging as a risk factor for development of diabetes and metabolic syndrome. Recently, it was shown in in-vitro cell culture experiments that hyperuricemia induces redox-dependent signaling and oxidative stress in adipocytes. By targeting levels of uric acid with febuxostat it is hypothesized that the levels of oxidative stress in adipose tissue (obtained by fat biopsy) will decrease.

Primary aims of the study are to determine whether febuxostat therapy in overweight or obese, diabetic patients with stage 3 Chronic Kidney Disease (CKD) and high serum uric acid levels

1. will affect adipose tissue concentrations of thiobarbituric acid reactive substance (TBARS), a marker of oxidative stress
2. will affect adipose tissue expression and concentrations of adiponectin; and
3. will affect urinary concentrations of transforming growth factor (TGF)- B1.

DETAILED DESCRIPTION:
Hyperuricemia is highly prevalent in the US population and commonly clusters with obesity and metabolic syndrome. It remains controversial whether this reflects an epiphenomenon or connotes a causal role of hyperuricemia in metabolic syndrome. If indeed hyperuricemia plays a causal role in metabolic syndrome, it would be expected that hyperuricemia will impact on the molecular signals that mediate the effects of adiposity on inflammation and insulin resistance.

Adipokines, the protein hormones produced by the adipocytes, serve as the signals for the effects of adipocytes on insulin resistance, dyslipidemia, hypertension, inflammation and atherosclerosis. Adipokines include tumor necrosis factor-α (TNF-α), interleukin-6 (IL-6), plasminogen activator inhibitor (PAI-1), leptin, angiotensinogen and adiponectin. In obesity, the production of TNF-α, IL-6, PAI-1, leptin and angiotensinogen increases whereas the production of adiponectin decreases. Increased expression of pro-inflammatory TNF-α and IL-6 and decreased expression of anti-inflammatory adiponectin by adipocytes results in insulin resistance and inflammation.

As oxidative stress in adipose tissue is considered to play a critical role in dysregulation of adipokines production in obesity and that hyperuricemia induces oxidative stress in adipocytes, it is hypothesized that hyperuricemia alters adipose tissue production of adipokines; therefore, febuxostat therapy will decrease hyperuricemia and thereby, have beneficial effects on adipokine production by adipose tissue; the favorable effects on adipokine production by febuxostat therapy will result in decrease in plasma levels of markers of inflammation; and as a result of the above, urinary markers of kidney disease will improve.

Chronic Kidney Disease (CKD) patients with type 2 diabetes will be studies because this population has a high prevalence of hyperuricemia and likely represents a target population which might benefit from reduction of uric acid levels.

This is a placebo-controlled, double-blinded, randomized controlled trial to examine the effects of uric acid lowering with oral febuxostat on adipokines and markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* BMI > 25 kg/m2
* type 2 diabetes
* serum uric acid ≥ 5.5 mg/dl in men and ≥ 4.6 mg/dl in women
* eGFR 30-60 mL/min/1.73m2

Exclusion Criteria:

* History of gout
* concurrent use of azathioprine, mercaptopurine, theophylline, allopurinol, thiazolidinediones or warfarin
* concurrent use of metformin
* current antibiotic therapy
* pregnant women
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasan Beddhu, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Beddhu S, Filipowicz R, Wang B, Wei G, Chen X, Roy AC, DuVall SL, Farrukh H, Habib AN, Bjordahl T, Simmons DL, Munger M, Stoddard G, Kohan DE, Greene T, Huang Y. A Randomized Controlled Trial of the Effects of Febuxostat Therapy on Adipokines and Markers of Kidney Fibrosis in Asymptomatic Hyperuricemic Patients With Diabetic Nephropathy. Can J Kidney Health Dis. 2016 Dec 5;3:2054358116675343. doi: 10.1177/2054358116675343. eCollection 2016. PMID 28270924

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Febuxostat | Placebo
Started | 40 | 40
Completed | 37 | 39
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Febuxostat | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (10) | 68 (11) | 68 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 24 | 28 | 52
Plasma Uric Acid Level [Mean (Standard Deviation); unit: milligram per deciliter] | 7.2 (1.5) | 7.1 (1.2) | 7.2 (1.4)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: milliliters per minute] | 52.2 (15.3) | 54.8 (19.0) | 53.5 (17.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Thiobarbituric Acid Reactive Substance (TBARS) Concentration in Adipose Tissue From Baseline to 24 Weeks
Description: The percent difference in thiobarbituric acid reactive substance (TBARS) concentration geometric mean values from baseline to 24 weeks was calculated for each arm
Time Frame: Baseline and 24 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: percent difference in geometric mean
Arm/Group | Febuxostat | Placebo
Number analyzed (Participants) | 37 | 39
percent difference in geometric mean | 34.0 [-26.3 to 143.4] | 44.6 [-19.3 to 159.2]
Statistical Analysis 1: Comparison: Febuxostat vs Placebo; Test type: Superiority or Other; p = 0.84, ANCOVA

2. Primary Outcome: Change in Adiponectin Concentration in Adipose Tissue From Baseline to 24 Weeks
Description: The percent difference in adiponectin concentration geometric mean values from baseline to 24 weeks was calculated for each arm
Time Frame: Baseline and 24 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: percent difference in geometric mean
Arm/Group | Febuxostat | Placebo
Number analyzed (Participants) | 37 | 39
percent difference in geometric mean | 2.3 [-23.4 to 36.7] | -4.1 [-27.7 to 27.4]
Statistical Analysis 1: Comparison: Febuxostat vs Placebo; Test type: Superiority or Other; p = 0.73, ANCOVA

3. Primary Outcome: Change in Urinary Concentrations of Transforming Growth Factor-beta1 (TGF-beta1) From Baseline to 24 Weeks
Description: The percent difference in TGF-beta1 concentration geometric mean values from baseline to 24 weeks was calculated for each arm
Time Frame: Baseline and 24 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: percent difference in geometric mean
Arm/Group | Febuxostat | Placebo
Number analyzed (Participants) | 37 | 39
percent difference in geometric mean | 29.8 [4.4 to 61.5] | 10.0 [-10.8 to 35.6]
Statistical Analysis 1: Comparison: Febuxostat vs Placebo; Test type: Superiority or Other; p = 0.23, ANCOVA

4. Secondary Outcome: Change in Tumor Necrosis Factor-α (TNF-α) Concentration in Plasma From Baseline to 24 Weeks
Description: The percent difference in plasma TNF-α concentration geometric mean values from baseline to 24 weeks was calculated for each arm
Time Frame: Baseline and 24 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: percent difference in geometric mean
Arm/Group | Febuxostat | Placebo
Number analyzed (Participants) | 37 | 39
percent difference in geometric mean | -9.9 [-30.6 to 16.8] | -7.4 [-28.3 to 19.7]
Statistical Analysis 1: Comparison: Febuxostat vs Placebo; Test type: Superiority or Other; p = 0.88, ANCOVA

5. Secondary Outcome: Change in Interleukin-6 (IL-6) Concentration in Plasma From Baseline to 24 Weeks
Description: The percent difference in plasma IL-6 concentration geometric mean values from baseline to 24 weeks was calculated for each arm
Time Frame: Baseline and 24 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: percent difference in geometric mean
Arm/Group | Febuxostat | Placebo
Number analyzed (Participants) | 37 | 39
percent difference in geometric mean | -24.0 [-35.3 to -10.7] | -9.5 [-22.7 to 6.1]
Statistical Analysis 1: Comparison: Febuxostat vs Placebo; Test type: Superiority or Other; p = 0.13, ANCOVA

6. Secondary Outcome: Change in High Sensitivity C-Reactive Protein (hsCRP) Concentration in Plasma From Baseline to 24 Weeks
Description: The percent difference in plasma hsCRP concentration geometric mean values from baseline to 24 weeks was calculated for each arm
Time Frame: Baseline and 24 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: percent difference in geometric mean
Arm/Group | Febuxostat | Placebo
Number analyzed (Participants) | 37 | 39
percent difference in geometric mean | 12.2 [-16.3 to 50.3] | -7.2 [-30.5 to 23.8]
Statistical Analysis 1: Comparison: Febuxostat vs Placebo; Test type: Superiority or Other; p = 0.35, ANCOVA

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: Details of adverse events experienced, particularly hospitalizations and emergency department visits obtained at each scheduled follow-up visit through week 24.
Arm/Group | Febuxostat | Placebo
Serious Adverse Events (participants affected / at risk) | 1/40 | 3/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Febuxostat (N=40) | Placebo (N=40)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ischemic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Flu-like Symptoms (General disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Aortic Valve Disease (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No